CLINICAL TRIAL: NCT01168011
Title: A Phase 1 Study To Assess The Tolerability, Pharmacokinetics and Clinical Activity of Rigosertib Administered Orally as Escalating Multiple Doses Twice or Three Times a Day up to 21 Days of a 21-Day Cycle in Patients With Advanced Cancer
Brief Title: Safety, Pharmacokinetics and Clinical Activity of Oral Rigosertib in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onconova 09-04; COMIRB # 10-0150 (Other: University of Colorado Cancer Center)
Record Dates: First submitted 2010-07-18; First posted 2010-07-22 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Solid Tumor
MeSH Terms: interventions — ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rigosertib (Experimental): Doses of rigosertib up to 700 mg twice a day or three times a day every day of 21-day cycles.
  Interventions: Drug: rigosertib

INTERVENTIONS:
Drug: rigosertib — Doses of rigosertib up to 700 mg twice a day or three times a day for 21 days of 21-day cycles. Treatment may continue until progression.
  Other Names: rigosertib sodium; ON 01910.Na

SUMMARY:
This is a phase 1 study in which 2 to 72 patients with advanced cancer will receive oral doses of rigosertib, a new investigational (unapproved) anti-cancer drug. The objective of the study is to determine the highest dose of drug that can be given safely. The study will start by testing a low dose. If this dose is safe, then, higher and higher doses will be tested as long as the previous lower dose was safe. Safety will be determined by looking for any side effects or unusual laboratory values. It is important to know the highest safe dose so that additional studies can be done. The drug will be given in the form of capsules twice or three times a day for 21 consecutive days of 21-day cycles.

DETAILED DESCRIPTION:
Patients will be initially enrolled in two-patient cohorts starting with a 70 mg bid dosing.

* In the absence of drug-related grade 2 or higher toxicity in the two patients treated for an entire 21-day first cycle, the next two patients will be receiving a dose escalated by 100% from prior dose.
* If drug-related grade 2 or higher toxicity is observed in at least one of the two patients treated for a full 21-day cycle, the cohort will be expanded in order to obtain 3 evaluable (treated for an entire 21-day first cycle) patients.
* If no dose limiting toxicity (DLT) is observed in the first three patients treated for an entire 21-day first cycle, then the next three patients will be enrolled at a dose level increased by approximately 50% from prior dose.
* If one DLT is observed in the first three patients treated for an entire 21-day first cycle, then the three next patients will be enrolled at the same dose level.
* If no more than one DLT is observed in the six patients treated for an entire 21-day cycle, then the next six patients will be administered a dose level increased by approximately 25% from prior dose.
* If two or more patients in any cohort experience DLT, then the maximum tolerated dose (MTD) will have been exceeded and no further dose escalation will occur. The MTD will be established as the immediate prior dosing level
* Identical rules will be applied to all cohorts of patients recruited to the study.
* A total of up to 24 patients may be treated at the MTD dose level in order to obtain data on the onset and severity of dysuria symptoms in approximately 12 patients including about 6 patients who will be treated with oral sodium bicarbonate at the time of treatment initiation (early treatment) and ~6 patients who will be treated with oral sodium bicarbonate at the time of symptom onset (late treatment). Alternating patients on a 1-to-1 basis by enrollment date will receive oral sodium bicarbonate as 650 mg tablets given twice daily with two 8-ounce glasses of water 1 hour after rigosertib administration, either at the time of study initiation (early treatment) or at the time of urinary symptom onset (late treatment).

Three additional cohorts will be treated with multiple escalating doses administered orally three time daily (TID) (140 mg, 280 mg and 420 mg) for 21 consecutive days of a 21-day cycle using identical rules as those described above (ie, starting with 2-patient cohorts at 140 mg dosing and expanding to 3-6 patient cohorts if at least 1 Grade 2 or higher drug-related toxicity is observed in 2-patient cohorts).

Up to 12 patients may be treated at the MTD level identified with TID dosing.

Prior to escalating to the next planned dose level, a designated Cohort Review Committee (CRC) consisting of the Principal Investigators (or their representatives), the Medical Monitor and the Sponsor's Medical Representative will review all available safety data over the 21 day duration of Course 1 for the previous cohort. Additional input may be provided from the study monitors, pharmacokinetic or toxicology specialists as required. The CRC also has to ability to recommend dose de-escalation for ON 01910.Na if warranted by the observed toxicity profile.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed solid tumor (leukemias and lymphomas excluded).
2. Malignancy that is incurable and for which standard (FDA approved or established standard clinical practice), curative, or palliative measures do not exist or are no longer effective.
3. ECOG performance status 2, 1 or 0.
4. Life expectancy greater than 6 months.
5. One or more measurable lesion(s) ("target lesion[s]"), that can be accurately measured in at least 1 dimension with longest diameter equal to or greater than 20 mm using conventional techniques (computed tomography [CT] scan or magnetic resonance imaging [MRI]) or equal to or greater than 10 mm with spiral CT scan.
6. If female, has a negative screening for pregnancy. Women of child-bearing potential and men must agree to use adequate contraception prior to study entry (hormonal or barrier method of birth control; abstinence) and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
7. Ability to understand the nature of the study and any hazards of participating in it, to communicate satisfactorily with the investigator, and to participate in, and comply with, the requirements of the entire study.
8. Willing to adhere to the prohibitions and restrictions specified in this protocol.
9. Patient must have signed an informed consent document.

Exclusion Criteria:

1. Recent major surgery (within the past 14 days).
2. Chemotherapy or dose of other potentially myelosuppressive treatment within 3 weeks prior to entering the study (6 weeks for nitrosoureas or mitomycin C).
3. Among patients with prior doxorubicin chemotherapy, only those with no more than a total cumulative dose of 450 mg/m2 of the drug.
4. Definitive radiotherapy (over 10 fractions and maximal area of hematopoietic active bone marrow treated was greater than 25%) within 4 weeks prior to entering the study.
5. Palliative radiotherapy (10 or less fractions) within 2 weeks prior to entering the study.
6. Residual adverse events (except alopecia, stable residual neuropathy, and residual hand, foot syndrome) and ascites requiring active medical management including paracentesis, peripheral bilateral edema, hyponatremia (serum value less than 130 Meq/L) due to previously administered agents, which have not recovered at grade 1 severity level or below before study entry.
7. Receiving any other investigational agents or concurrent chemotherapy, radiotherapy, hormonal treatments, bone marrow transplantation, or immunotherapy while on study. Exceptions are long-term hormonals for prostate (e.g. goserelin) and octreotide for neuroendocrine malignancies.
8. Previous bone marrow transplant.
9. Known brain metastases, except brain metastases that have been previously removed or irradiated and currently have no clinical impact.
10. History of allergic reactions attributed to compounds of similar chemical or biologic composition to ON 01910.Na.
11. Uncontrolled intercurrent illness.
12. Hgb less than 9 gm/dL (must not require transfusional support but erythropoietin therapy is permitted).
13. WBC less than 4,000/microliter.
14. Absolute neutrophil count less than 1,500/microliter.
15. Platelets less than or equal to 100,000/microliter.
16. Total bilirubin greater than 1.5 times institutional upper normal limit.
17. AST(SGOT)/ALT(SGPT) equal to or greater than 2.5 x institutional upper normal limit. (If liver function abnormalities are due to metastatic disease, patients are eligible provided the transaminases are < 5 times institutional upper normal limit.).
18. Serum creatinine greater than 2 times upper limit of institutional normal value.
19. Pregnant and nursing women.
20. HIV-1 positive patients receiving combination anti-retroviral therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 2 years
  Adverse events (AEs) will be regarded as treatment emergent signs and symptoms (TESS) if they started on or after the date and time of administration of the first dose of study drug, or if they were present prior to the administration of the first dose of study drug and increased in severity during the study. Adverse events include clinical laboratory parameters (e.g., Hematology Panel and Serum Chemistry Panel). Other safety parameters include vital signs, physical examination findings, concomitant medications, and drug exposure.

SECONDARY OUTCOMES:
Concentration of ON 01910.Na in plasma | 2 years
  The concentration of ON 01910.Na in plasma at various times after administration will be used to derive the following PK parameters for ON 01910.Na using model-independent analysis as appropriate for the data: Tmax, Cmax, t½, AUC0-t, AUC 0-α, CL, and Vss.
Measurement of tumor size | 2 years
  Tumor response rates will be evaluated for each patient using RECIST criteria.
Concentration of ON 01910.Na in Urine | 1 years
  Urine PK samples to determine ON 01910.Na urinary concentrations will be collected on Day 1 and Day 21 of the first cycle, and on Day 15 of the second cycle in all patients and will include the predose void volume and a 24-hr post-dose urine collection over the 0-4 hr, 4-8 hr, and 8-24 hr intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Jimeno, MD, PhD, Principal Investigator — University of Colorado at Denver Health and Sciences
Locations (1):
- University of Colorado at Denver Health and Sciences, Denver, Colorado, United States

REFERENCES:
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.
- See also: Clinical Trials at University of Colorado Hospital — http://www.uch.edu/conditions/cancer/research/research_trials/index.aspx